CLINICAL TRIAL: NCT00855387
Title: Surgical Complications Dramatically Influence Overall Cost of Major Surgical Procedures
Brief Title: Severe Complications Triplicate the Costs of Major Surgical Procedures
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: R. Vonlanthen/Dr. med., University Hospital of Zurich
Other Study IDs: StV 5-2009
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Major Surgical Procedures
Keywords: Clinical outcome (complications), in-hospital costs; The influence and impact of postoperative complications on in-hospital costs
MeSH Terms: interventions — Pancreatic Hormones; Liver Extracts; Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Costs: Patients collected consecutively for undergoing major surgical procedures(liver, bile duct, pancreas, small bowel, colo-rectal, gastric bypass resections).
  Interventions: Other: No additional intervention than the intended major surgery in pancreas, liver, colorectal, gastric bypass and small bowel

INTERVENTIONS:
Other: No additional intervention than the intended major surgery in pancreas, liver, colorectal, gastric bypass and small bowel — No additional intervention than the intended major surgery (liver, bile duct, pancreas, colorectal, gastric bypass and small bowel resections) comparing with costs

SUMMARY:
The purpose of this study is to prospectively assess the impact of surgical quality on the overall cost of major surgical procedures using the incidence and severity of complications as surrogate markers of quality.

DETAILED DESCRIPTION:
To prospectively assess the impact of surgical quality on the overall cost of major surgical procedures using the incidence and severity of complications as surrogate markers of quality

ELIGIBILITY:
Inclusion Criteria:

* Undergoing major surgery (liver, bile duct, pancreas, colorectal, gastric bypass and small bowel resections)

Exclusion Criteria:

* Missing data of in-hospital costs
* Mortality

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort study with 1235 patients including consecutive patients undergoing major surgery (liver, bile duct, pancreas, colorectal, gastric bypass and small bowel resections) in a single tertiary care center
Sampling Method: Non-Probability Sample
Enrollment: 1235 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Clinical outcome (complications) In-hospital Costs | inhospital; peri-operative

CONTACTS AND LOCATIONS:
Overall Officials: René Vonlanthen, Dr. med., Principal Investigator — Department of Visceral and Transplantation Surgery
Locations (1):
- University Hospital of Zurich, Department of Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Vonlanthen R, Slankamenac K, Breitenstein S, Puhan MA, Muller MK, Hahnloser D, Hauri D, Graf R, Clavien PA. The impact of complications on costs of major surgical procedures: a cost analysis of 1200 patients. Ann Surg. 2011 Dec;254(6):907-13. doi: 10.1097/SLA.0b013e31821d4a43. PMID 21562405